CLINICAL TRIAL: NCT00393731
Title: A Randomized, Control Trial for Preinduction Cervical Ripening
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Michael Lucas, M.D., The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-04-008
Record Dates: First submitted 2006-10-26; First posted 2006-10-30 (Estimated); Last update posted 2008-01-16 (Estimated); Status verified 2008-01

CONDITIONS: Labor, Induced
Keywords: labor; induction; misoprostol; oxytocin
MeSH Terms: interventions — Misoprostol; Oxytocin

INTERVENTIONS:
Drug: Misoprostol
Drug: oxytocin

SUMMARY:
The goal of this study is to compare the vaginal delivery rates in women undergoing induction of labor with an unripe cervix between oxytocin induction alone and preinduction cervical ripening with prostaglandin El (misoprostol). Secondary goals are to measure and compare the time intervals to delivery between the two methods.

ELIGIBILITY:
Inclusion Criteria:

* Women that are hospitalized for induction of labor that have a Bishop's score <5
* singleton gestation
* cephalic presentation
* 24 weeks gestational age

Exclusion Criteria:

* Prior uterine surgery
* malpresentation
* placenta previa or abruption
* clinically suspected or diagnosed intra amniotic infection
* genital HSV infection
* multiple gestation
* premature rupture of the membranes
* active labor
* maternal/fetal conditions that may preclude labor induction in the opinion of the investigators

Sex: Female
Age Groups: Child, Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2004-01; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Vaginal Delivery rates

SECONDARY OUTCOMES:
Time interval to delivery

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lucas, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Lyndon B. Johnson Hospital, Houston, Texas, United States